CLINICAL TRIAL: NCT00656578
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate Efficacy and Safety of a Single Intraoperative Administration of 4975 in Patients Undergoing Unilateral Transpositional First Metatarsal Osteotomy for the Correction of Hallux Valgus Deformity
Brief Title: Efficacy and Safety Study of 4975 to Manage Pain of Bunionectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Anesiva, Inc. (Industry)
Responsible Party: Denise Sharp - CRA, Anesiva, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 114-08P
Record Dates: First submitted 2008-04-07; First posted 2008-04-11 (Estimated); Last update posted 2009-05-04 (Estimated); Status verified 2009-05

CONDITIONS: Pain
Keywords: Foot; Bunion; Bunionectomy; Hallux Valgus Deformity; Surgery for Transpositional first metatarsal osteotomy - Bunionectomy
MeSH Terms: conditions — Pain; Bunion | interventions — 7-propyltheophylline dopamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 4975
  Interventions: Drug: 4975
- 2 (Placebo Comparator): Drug, Single dose, solution
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 4975 — Single dose, solution
  Arms: 1
Drug: Placebo — Single dose, solution
  Arms: 2

SUMMARY:
The primary purpose of this study is to compare the analgesic efficacy of a single intraoperative administration of 4975 vs. Placebo in the management of acute postoperative pain in patients undergoing bunionectomy.

Secondary objective of this study is to evaluate the safety and tolerability of a single intraoperative administration of 4975.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled, parallel-group study conducted in the US. A dose of 4975 will be evaluated against placebo in patients undergoing bunionectomy. Upon enrollment, patients will be randomized in a 1:1 ratio to receive either 4975 or placebo.

After the surgery, patients will be admitted to the clinical study site, where trained study personnel will monitor them for up to 48 hours. While at the clinical study site, patients will undergo safety and efficacy assessments. After discharge, patients will report pain severity daily through Day 14 via an interactive voice response system (IVRS). Also, safety and patient-reported outcome assessments will be performed at the Day 14 (Week 2) and Day 28 (Week 4) clinic visits.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 years and older.
* Planning to undergo unilateral transpositional first metatarsal osteotomy for correction of Hallux Valgus Deformity (referred to as bunionectomy in this protocol).

Exclusion Criteria:

* Use of certain medications or having a medical condition that in the investigator's opinion could adversely impact the patient's participation or safety, conduct of the study, or interfere with the pain assessments.
* Diabetes mellitus with a known HbA1C > 9.5 or a history of prolonged uncontrolled diabetes.
* Participated in another clinical trial or used an investigational product within 30 days prior to the planned bunionectomy surgery, or is scheduled to receive an investigational product other than 4975 while participating in the study.
* Previously participated in a clinical study with 4975.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2008-03; Primary Completion 2008-08 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Evaluate efficacy of a single intraoperative administration of 4975 in the management of acute postoperative pain in patients undergoing bunionectomy | Prospective

SECONDARY OUTCOMES:
Evaluate safety and tolerability of a single intraoperative administration of 4975 | Prospective

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Foot and Ankle Institute, Bakersfield, California
  - Crossroads Research, Inc., Owings Mills, Maryland
  - Scirex Research Center, Austin, Texas
  - San Antonio Podiatry Associates, PC, San Antonio, Texas
  - Hill Country Sports Medicine of Podiatric Surgery, San Marcos, Texas
  - Scirex Research Center, Salt Lake City, Utah

REFERENCES:
- See also: Anesiva, Inc. Home page — http://www.anesiva.com/wt/page/pipeline
- See also: 4975 Product Information — http://www.anesiva.com/wt/page/adlea